CLINICAL TRIAL: NCT07173023
Title: A Comparative Study of Endoscopic Choanal Canalization and Mitomycin C Application vs Endoscopic Crossover Flap Technique
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ebram Hamdy Dawood Zaky, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: endoscopic choanal repair
Record Dates: First submitted 2025-09-04; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Choanal Atresia
MeSH Terms: conditions — Choanal Atresia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Transnasal Puncture with Mitomycin C application (Active Comparator): * Performed under general anesthesia.
  * Nasal cavities decongested with oxymetazoline.
  * Atretic plate perforated using serial dilators under direct visualization.
  * Additional removal of bony/membranous tissue including the posterior nasal septum as possible.
  * Topical mitomycin C (0.5 mg/mL) applied to the edges of the newly created choana for 2 minutes using cotton pledget in a transparent tube , followed by irrigation with saline.
  * syndromatic patients and patients requiring less time UGA will be included in this group
  Interventions: Procedure: Transnasal Puncture with Mitomycin C application
- Group 2: Endoscopic Crossover Flap Repair (Active Comparator): * Performed under general anesthesia using a 0° 4 mm endoscope.
  * Elevation of mucosal crossover flaps to cover exposed bone following resection of the atretic plate where one flap is inferiorly based and the other is superiorly based.
  * Precise removal of the posterior vomer and lateral bony plates as needed using cold steel instruments and possible nasal drill.
  * Flaps will be repositioned to minimize exposed bone and promote mucosal healing preventing restenosis.
  Interventions: Procedure: Endoscopic Crossover Flap Repair

INTERVENTIONS:
Procedure: Transnasal Puncture with Mitomycin C application — * Performed under general anesthesia.
  * Nasal cavities decongested with oxymetazoline.
  * Atretic plate perforated using serial dilators under direct visualization.
  * Additional removal of bony/membranous tissue including the posterior nasal septum as possible.
  * Topical mitomycin C (0.5 mg/mL) applied to the edges of the newly created choana for 2 minutes using cotton pledget in a transparent tube , followed by irrigation with saline.
  * syndromatic patients and patients requiring less time UGA will be included in this group
  Arms: Group 1: Transnasal Puncture with Mitomycin C application
Procedure: Endoscopic Crossover Flap Repair — * Performed under general anesthesia using a 0° 4 mm endoscope.
  * Elevation of mucosal crossover flaps to cover exposed bone following resection of the atretic plate where one flap is inferiorly based and the other is superiorly based.
  * Precise removal of the posterior vomer and lateral bony plates as needed using cold steel instruments and possible nasal drill.
  * Flaps will be repositioned to minimize exposed bone and promote mucosal healing preventing restenosis.
  Arms: Group 2: Endoscopic Crossover Flap Repair

SUMMARY:
determine the optimal surgical strategy for achieving

1. long-term outcomes
2. minimizing complications
3. improving outcomes in CCA patients

DETAILED DESCRIPTION:
Congenital choanal atresia (CCA) is a relatively common congenital nasal anomaly, characterized by the failure of canalization of the posterior nasal passage during embryological development, which normally occurs between the 4th and 11th weeks of gestation[1]. This developmental failure results in an obstruction-either bony, membranous, or mixed-at the posterior nasal aperture, leading to compromised nasal airflow[1]. Failure of canalization results in a persistent bucco-pharyngeal membrane or naso-buccal blockage, either bony or membranous in structure CCA affects approximately 1 in 5,000 to 8,000 live births, with a slight female predominance (twice as common in females).

Two-thirds of cases are unilateral, while one-third are bilateral. Risk factors include twin pregnancies, chromosomal anomalies, and antithyroid treatment during pregnancy.

Bilateral CCA is a neonatal emergency as infants are obligatory nasal breathing , leading to severe respiratory distress, cyclical cyanosis, and feeding difficulties immediately after birth.

Diagnosis is suspected when a soft catheter cannot pass through the nose and confirmed by CT scan.

Nearly half of the affected neonates have additional syndromic anomalies, such as CHARGE syndrome, highlighting the need for comprehensive evaluation The main goal of surgery is to create an patent nasal airway; techniques have evolved from the traditional transpalatal approach to minimally invasive transnasal endoscopic methods.

The transpalatal approach is less favored now due to higher risks of complications such as palatal fistulas and dental deformities.

Endoscopic transnasal techniques are now preferred as they offer better visualization, less morbidity, minimal blood loss, and avoidance palatal growth disturbance.

Simple transnasal endoscopic canalization is technically easy but may have higher rates of restenosis compared to more advanced techniques using mucosal flaps.

Using mucosal flaps in endoscopic surgery can reduce scar tissue and restenosis by providing mucosal coverage and minimizing granulation tissue formation.

Stents are sometimes used for 6-8 weeks, but their necessity and benefits remain debated, with some protocols avoiding stenting altogether.

Topical mitomycin C is used by some surgeons to prevent scar formation, but its effectiveness is still controversial.

There is a need for prospective randomized studies to determine the most suitable approach for long-term success and fewer complications in CCA patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-72 months at enrollment.
* Diagnosis of congenital choanal atresia (unilateral or bilateral) confirmed by nasal endoscopy and CT imaging.
* Patients presenting with clinical symptoms (e.g., nasal obstruction, respiratory distress, feeding difficulties) or requiring surgical intervention.
* Guardians willing to provide informed consent and comply with follow-up.

Exclusion Criteria:

* Acquired (non-congenital) choanal atresia.
* Previous surgical intervention for choanal atresia.
* Significant comorbidities contraindicating surgery (e.g., unstable cardiopulmonary status).
* Incomplete medical records or anticipated inability to complete follow-up.

Ages: 0 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Rate of restenosis at 12 months postoperatively, defined as symptomatic obstruction confirmed by endoscopy and/or CT scan. | 12 months postoperatively
  Rate of restenosis at 12 months postoperatively, defined as symptomatic obstruction confirmed by endoscopy and/or CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: ebram hamdy dawood, resident doctor, Principal Investigator — Assiut University; Moustafa omar Mohammed Ali, lecturer, Study Director — Assiut University; ezzat mohammed saleh, professor doctor, Study Director — Assiut University

REFERENCES:
- [Background] Al-khatib T, Haneef SH, Alhusaini OA, et al. Transnasal puncture technique vs endoscopic transnasal choanal atresia repair. J Otolaryngol ENT Res. 2019;11(2):124?127. DOI: 10.15406/joentr.2019.11.00421
- [Background] Deutsch E, Kaufman M, Eilon A. Transnasal endoscopic management of choanal atresia. Int J Pediatr Otorhinolaryngol. 1997 May 4;40(1):19-26. doi: 10.1016/s0165-5876(96)01486-3. PMID 9184974
- [Background] Bajin MD, Onay O, Gunaydin RO, Unal OF, Yucel OT, Akyol U, Aydin C. Endonasal choanal atresia repair; evaluating the surgical results of 58 cases. Turk J Pediatr. 2021;63(1):136-140. doi: 10.24953/turkjped.2021.01.016. PMID 33686836
- [Background] Llorente JL, Lopez F, Morato M, Suarez V, Coca A, Suarez C. Endoscopic treatment of choanal atresia. Acta Otorrinolaringol Esp. 2013 Nov-Dec;64(6):389-95. doi: 10.1016/j.otorri.2013.05.001. Epub 2013 Jul 27. English, Spanish. PMID 23896489
- [Background] Stamm AC, Pignatari SS. Nasal septal cross-over flap technique: a choanal atresia micro-endoscopic surgical repair. Am J Rhinol. 2001 Mar-Apr;15(2):143-8. doi: 10.2500/105065801781543718. PMID 11345154